CLINICAL TRIAL: NCT04510545
Title: Real-Time Artificial Intelligence Aided Diagnosis of Colorectal Polyps During Colonoscopy: A Clinical Trial With the EndoBRAIN Technology
Brief Title: Computer Aided Diagnosis of Colorectal Polyps
Acronym: EndoBrain
Status: Completed | Type: Observational
Sponsor: King's College Hospital NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 260047
Record Dates: First submitted 2019-09-24; First posted 2020-08-12 (Actual); Last update posted 2022-01-31 (Actual); Status verified 2022-01

CONDITIONS: Colonic Polyp; Colorectal Cancer
MeSH Terms: conditions — Colonic Polyps; Colorectal Neoplasms | interventions — Diagnosis, Computer-Assisted

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Treatment Group: All patients will undergo CAD of any diminutive polyps found in the rectosigmoid on colonoscopy
  Interventions: Diagnostic Test: Endobrain, Computer Aided Diagnosis (CAD)

INTERVENTIONS:
Diagnostic Test: Endobrain, Computer Aided Diagnosis (CAD) — Artificial intelligence

SUMMARY:
The purpose of this study is to assess whether computer aided technology (CAD) can help in the diagnosis of polyps found the bowel compared with visual inspection alone and therefore whether it is beneficial in helping clinicians to decide whether to remove a polyp or not. Presently, most endoscopists remove all polyps found and send them to the laboratory for testing. The number of colonoscopies is increasing, meaning that more polyps are detected and removed. This comes at a significant cost to the health service and increases the time taken to complete a colonoscopy.

DETAILED DESCRIPTION:
Removing precancerous polyps from the bowel during a colonoscopy (camera test) is the cornerstone of colorectal cancer screening and prevents polyps developing into bowel cancer. Most polyps develop in the rectosigmoid colon (lower part of the bowel). Many polyps never grow into cancer and it can be difficult for the clinicians performing the procedure (endoscopists) to tell which ones are precancerous. This means many polyps are removed unnecessarily, with a considerable waste of resources.

A recent preliminary study indicates a novel artificial intelligence system (EndoBRAIN) for computer-aided diagnosis may be able to distinguish different types of polyps during colonoscopy and therefore help doctors decide which polyps to remove. This study aims to compare the in accuracy of artificial intelligence against the endoscopist's assessment for diagnosis of diminutive (<5mm) polyps in the lower colon.

Patients who are age 18 years or older who undergo colonoscopy for any indication at the participating clinical centres and are diagnosed with diminutive rectosigmoid polyps are eligible for study enrolment. For each detected polyp in the rectosigmoid colon, endoscopists will assess the polyp type using standard colonoscopies (cameras) and then with the use of the EndoBRAIN technology.

The polyps will be removed and sent to the laboratory for testing. The difference between clinician diagnosis and EndoBRAIN diagnosis will be compared with the laboratory findings. We hypothesize that the EndoBRAIN technology provides a superior accuracy in identifying precancerous rectosigmoid polyps, compared to endoscopist's own prediction with a standard colonoscope.

If the trial confirms the superior accuracy of the EndoBRAIN system, polyps classified as non-cancerous with the EndoBRAIN system no longer need to be removed, meaning a large gain for patients and society, due to significantly less polypectomies and pathology reviews.

ELIGIBILITY:
Inclusion Criteria:

* Individuals 18 years or older who are scheduled for screening, surveillance, diagnostic, or therapeutic colonoscopy at at King's College Hospital with diminutive rectosigmoid polyps.

Exclusion Criteria:

* Diminutive polyps with known histology
* Inflammatory bowel disease
* Polyposis syndrome (e.g., familial adenomatous polyposis, serrated polyposis)
* History of chemotherapy or radiation therapy for colorectal lesions
* Inability to undergo polypectomy (e.g. intake of anticoagulants, comorbidities, or patient refusal)
* Pregnancy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Any patient 18 years or older scheduled for screening, surveillance, diagnostic, or therapeutic colonoscopy at King's College Hospital with diminutive rectosigmoid polyps.
Sampling Method: Non-Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-05-05 (Actual); Study Completion 2021-05-05 (Actual)

PRIMARY OUTCOMES:
True positive adenoma detection rate | 6 months
  True positive adenoma detection rate with visual inspection versus true positive adenoma detection rate with visual inspection plus CAD

SECONDARY OUTCOMES:
True negative adenoma detection rate | 6 months
  True negative adenoma detection rate with visual inspection versus true negative adenoma detection rate with visual inspection plus CAD
To estimate the sensitivity, specificity, of visual inspection and the use of the EndoBRAIN CAD technology | 6 months
  To estimate the sensitivity, specificity, of visual inspection and the use of the EndoBRAIN CAD technology
To estimate the positive predictive value [PPV], and NPV of the combination of visual inspection and the use of the EndoBRAIN CAD technology | 6 months
  To estimate the positive predictive value [PPV], and NPV of the combination of visual inspection and the use of the EndoBRAIN CAD technology
To estimate the percentage of diminutive colorectal polyps from which endocytoscopic images can be successfully captured (acquisition rate). | 6 months
  To estimate the percentage of diminutive colorectal polyps from which endocytoscopic images can be successfully captured (acquisition rate).
To estimate the rate of high-confidence diagnosis with EndoBRAIN as compared to visual polyp inspection alone. | 6 months
  To estimate the rate of high-confidence diagnosis with EndoBRAIN as compared to visual polyp inspection alone.
Time of colonoscopy | during procedure
  Time of colonoscopy to be recorded.
Complications | 6 months
  complications to be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- King's College Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
The IPD will be kept within the research team.